CLINICAL TRIAL: NCT04867161
Title: Superinfection and Hyperinflammatory Phenotype in COVID-19 (Coronavirus Disease 2019) Pneumonia Patients (SUPER-HI) - Prospective Observational Study
Brief Title: Superinfection and Hyperinflammatory Phenotype in COVID-19 (Coronavirus Disease 2019) Pneumonia Patients
Acronym: SUPER-HI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Jan Malaska, Principal investigator, Brno University Hospital
Other Study IDs: 146/20
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: COVID-19 Pneumonia; Superinfection Lung
Keywords: COVID-19; superinfection; inflammatory markers
MeSH Terms: conditions — COVID-19; Superinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum samples and bronchoalveolar fluid samples are stored in aliquots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with COVID-19 pneumonia without superinfection: Patients with confirmed COVID-19 pneumonia not fulfilling criteria for diagnosis HAP/VAP (International ERS/ESICM/ESCMID/ALAT guidelines for the management of hospital-acquired pneumonia and ventilator-associated pneumonia )
  Interventions: Diagnostic Test: Inflammatory markers sampling
- Patients with COVID-19 pneumonia with superinfection: Patients with confirmed COVID-19 pneumonia fulfilling criteria for diagnosis HAP/VAP (International ERS/ESICM/ESCMID/ALAT guidelines for the management of hospital-acquired pneumonia and ventilator-associated pneumonia )
  Interventions: Diagnostic Test: Inflammatory markers sampling

INTERVENTIONS:
Diagnostic Test: Inflammatory markers sampling — Laboratory sampling:
  Haematology: complete blood count, reticulocytes, IFP, PT, aPTT, fibrinogen, D-dimer Biochemical profile: urea, creatinine, bilirubin, ALT, AST, GGT, CK, LD, ferritin, troponin Inflammation markers IL-6, PCT (procalcitonin), CRP (C-reactive protein), PSP (presepsin)
  BALF (bronchoalveolar lavage fluid) processing protocol:
  1. microbiology: microscopic examination, standard cultivation test
  2. biochemistry: albumin, total protein
  3. Pathology: cytology
  4. PCR:
  a. Multiplex PCR b. SARS-CoV-2 RNA load

SUMMARY:
Patients suffering from COVID-19 (Coronavirus Disease 2019) pneumonia are prone to bacterial and mycotic superinfection. According to existing evidence, the prevalence of superinfection is about 8% to 14% (95% CI 5-26%). However, the percentage of patients treated for superinfection is as high as 80%. There can be multiple reasons for this difference.

DETAILED DESCRIPTION:
The inflammatory markers, such as C-reactive protein (CRP), procalcitonin (PCT), presepsin (PSP), interleukin-6 (IL-6) frequently used as diagnostic tools in COVID-19 (Coronavirus Disease 2019), are usually increased in these patients. This increase is a result of activation of systemic inflammatory cascade, part of COVID-19 pathophysiologic pathway. This can escalate to state known as COVID-19 associated hyperinflamation (COV-HI). In addition, current diagnostic tools for diagnosing HAP/VAP (hospital-acquired pneumonia and ventilator-associated pneumonia) are often limited in patients with COVID-19 pneumonia. The current method of choice for superinfection diagnosing is BAL (Bronchoalveolar Lavage). The COV-HI phenotype (COV-HI: CRP > 150 mg/L, or doubling within 24 h from greater than 50 mg/L, or ferritin concentration > 1500 ug/L) is associated with significantly worse course of illness and higher mortality rates. These inflammatory markers may be used preferentially as prognostication tools, not bacterial superinfection markers. The intention of this project is to investigate the role of currently used inflammatory biomarkers. Or eventually, to discover new parameters associated with superinfection proven by BAL.

ELIGIBILITY:
Inclusion Criteria:

1. admission on ICU
2. age more than 18 years
3. COVID-19 pneumonia criteria fulfilled

Exclusion Criteria: none

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 diagnostics:
  PCR test from nasopharyngeal swab or tracheal aspirate plus Chest X-ray/Computer tomography signs of pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers dynamics in participants with superinfection in COVID-19 pneumonia | 28 days
  To investigate the role of inflammatory markers (CRP, PCP, PSP, IL-6) as diagnostic tools for superinfection in COVID-19 pneumonia patients.

SECONDARY OUTCOMES:
Mortality from any cause | 28, 60, 90, 180, 360 days
  To assess the association between hyperinflammatory phenotype and course of illness and mortality rates in COVID-19 pneumonia patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Maláska, Principal Investigator — Brno University Hospital
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rawson TM, Moore LSP, Zhu N, Ranganathan N, Skolimowska K, Gilchrist M, Satta G, Cooke G, Holmes A. Bacterial and Fungal Coinfection in Individuals With Coronavirus: A Rapid Review To Support COVID-19 Antimicrobial Prescribing. Clin Infect Dis. 2020 Dec 3;71(9):2459-2468. doi: 10.1093/cid/ciaa530. PMID 32358954
- [Background] Lansbury L, Lim B, Baskaran V, Lim WS. Co-infections in people with COVID-19: a systematic review and meta-analysis. J Infect. 2020 Aug;81(2):266-275. doi: 10.1016/j.jinf.2020.05.046. Epub 2020 May 27. PMID 32473235
- [Background] Keddie S, Ziff O, Chou MKL, Taylor RL, Heslegrave A, Garr E, Lakdawala N, Church A, Ludwig D, Manson J, Scully M, Nastouli E, Chapman MD, Hart M, Lunn MP. Laboratory biomarkers associated with COVID-19 severity and management. Clin Immunol. 2020 Dec;221:108614. doi: 10.1016/j.clim.2020.108614. Epub 2020 Oct 22. PMID 33153974
- [Background] Manson JJ, Crooks C, Naja M, Ledlie A, Goulden B, Liddle T, Khan E, Mehta P, Martin-Gutierrez L, Waddington KE, Robinson GA, Ribeiro Santos L, McLoughlin E, Snell A, Adeney C, Schim van der Loeff I, Baker KF, Duncan CJA, Hanrath AT, Lendrem BC, De Soyza A, Peng J, J'Bari H, Greenwood M, Hawkins E, Peckham H, Marks M, Rampling T, Luintel A, Williams B, Brown M, Singer M, West J, Jury EC, Collin M, Tattersall RS. COVID-19-associated hyperinflammation and escalation of patient care: a retrospective longitudinal cohort study. Lancet Rheumatol. 2020 Oct;2(10):e594-e602. doi: 10.1016/S2665-9913(20)30275-7. Epub 2020 Aug 21. PMID 32864628
- [Background] WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection. A minimal common outcome measure set for COVID-19 clinical research. Lancet Infect Dis. 2020 Aug;20(8):e192-e197. doi: 10.1016/S1473-3099(20)30483-7. Epub 2020 Jun 12. PMID 32539990